CLINICAL TRIAL: NCT00310037
Title: A Randomized Phase II Trial of Maintenance vs Consolidation Bortezomib Therapy Following Aggressive Chemo-Immunotherapy and Autologous Stem Cell Transplant for Previously Untreated Mantle Cell Lymphoma
Brief Title: Bortezomib After Combination Chemotherapy, Rituximab, and an Autologous Stem Cell Transplant in Treating Patients With Mantle Cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CALGB-50403; CDR0000466167 (Other: NCI Physician Data Query)
Record Dates: First submitted 2006-03-29; First posted 2006-04-03 (Estimated); Results first posted 2018-07-31 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Mantle Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A maintenance therapy (Experimental): Patients receive bortezomib 1.6 mg/m^2 IV on days 1, 8, 15, and 22 once daily for 4 weeks. There will be a 4 week rest period. One cycle is a total of 8 weeks. A total of 10 cycles of bortezomib will be given in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: bortezomib
- Arm B consolidation therapy (Experimental): Patients receive bortezomib 1.3 mg/m^2 IV on days 1, 4, 8, and 11 once daily for 3 weeks. One cycle is a total of 3 weeks. A total of 4 cycles of bortezomib will be given in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: bortezomib

INTERVENTIONS:
Drug: bortezomib — Given IV

SUMMARY:
This randomized phase II trial studies how well bortezomib works when given after combination chemotherapy, rituximab, and an autologous stem cell transplant in treating patients with mantle cell lymphoma. Bortezomib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) together with an autologous stem cell transplant may allow more chemotherapy to be given so that more cancer cells are killed. Monoclonal antibodies, such as rituximab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. Giving bortezomib after combination chemotherapy, monoclonal antibody therapy, and an autologous stem cell transplant may kill any remaining cancer cells or keep the cancer from coming back.

DETAILED DESCRIPTION:
Objectives

Primary Objective:

To determine the 18-month progression-free survival (PFS) in patients with previously untreated mantle cell lymphoma who are treated with aggressive chemo-immunotherapy and autologous stem cell transplant followed by randomization to either maintenance or consolidation bortezomib therapy

Secondary Objectives:

* To determine the toxicity profiles of maintenance and consolidation bortezomib by evaluating the number of patients able to complete all maintenance or consolidation therapy
* To determine the complete response rate to intensive chemo-immunotherapy plus maintenance or consolidation bortezomib
* To determine time to progression and overall survival using these two treatment regimens

Correlative/Other Pre-Specified Objectives:

* To determine the importance of p53 mutation or deletion on patient outcome with respect to CR rate, PFS, and OS
* To determine the importance of Ki67, cyclin D1, phosphohistone 3, p27, p21, p16, and PARP p85 expression in pre-treatment tumor biopsies with respect to CR rate, PFS, and OS
* To determine the relationship between proliferation signature and clinical outcome using quantitative real-time RT-PCR
* To evaluate the importance of quantitative cyclin D1 expression and expression of cyclin D1 isoforms in predicting clinical outcome using quantitative real-time RT-PCR
* To evaluate the prognostic significance of microRNAs in mantle cell lymphoma using microRNA arras
* To explore the correlation of selected microRNA polymorphisms with gene target expression with clinical outcomes such as response, PFS, and OS
* To determine changes in gene expression profile from diagnosis to relapse samples to identify genes differentially silenced or over-expressed with disease recurrence
* To determine the importance of early PCR negativity (following Treatment 2) using bcl-1/IgH junction and/or IgH chain gene rearrangement with respect to maintained PFS and the success of maintenance or consolidation therapy to converting patients to PCR negative status

OUTLINE OF INTERVENTIONS:

CHEMOIMMUNOTHERAPY: Patients receive chemoimmunotherapy comprising rituximab* intravenously (IV) over 4-6 hours on day 1, methotrexate (MTX) IV over 4 hours on day 2, cyclophosphamide IV over 2 hours, doxorubicin hydrochloride IV, and vincristine sulfate IV on day 3, and prednisone orally (PO) on days 3-7. Beginning 24 hours after completion of MTX, patients receive leucovorin calcium IV every 6 hours until blood levels of MTX are in a safe range. Patients also receive filgrastim (G-CSF) subcutaneously (SC) once daily (QD) beginning on day 3 and continuing until blood counts recover. Beginning no sooner than day 22, but no later that day 29 of the first course, patients receive a second course of chemoimmunotherapy as above. Patients with > 15% persistent bone marrow involvement may receive a third course of chemoimmunotherapy. Patients are restaged and those with progressive disease are removed from therapy.

NOTE: *During the first course of chemoimmunotherapy, patients receive rituximab only if the number of circulating mantle cells is =< 10,000/mm^3, otherwise, rituximab is omitted during the first course of chemoimmunotherapy.

HIGH-DOSE CONSOLIDATION CHEMOIMMUNOTHERAPY AND PERIPHERAL BLOOD STEM CELL (PBSC) COLLECTION: Approximately 4 weeks after completion of chemoimmunotherapy, patients receive high-dose consolidation chemoimmunotherapy comprising cytarabine IV over 2 hours and etoposide phosphate IV continuously on days 1-4, and rituximab IV over 4-6 hours on days 5 and 12 OR 6 and 13. Beginning on day 14 and continuing until completion of PBSC collection, patients receive G-CSF SC QD. Once blood counts recover, patients undergo 1-3 leukapheresis procedures for collection of PBSCs on days 22-25.

HIGH-DOSE CHEMOTHERAPY AND AUTOLOGOUS PBSC TRANSPLANTATION (PBSCT): Beginning 4-6 weeks after completion of leukapheresis, patients receive carmustine IV over 2 hours on day -6, etoposide phosphate IV over 4 hours on day -4, and cyclophosphamide IV over 2 hours on day -2. Patients undergo autologous PBSCT on day 0. Patients also receive G-CSF SC QD beginning on day 4 and continuing until blood counts recover.

POST-TRANSPLANTATION IMMUNOTHERAPY: Approximately 5 weeks after autologous PBSCT, patients receive rituximab IV over 4-6 hours once weekly for 2 weeks. Approximately 4 weeks after completion of post-transplantation immunotherapy, patients proceed to maintenance therapy or consolidation therapy with bortezomib as described in the Arms section.

After completion of study treatment, patients are followed every 2 months for 2 years, every 6 months for 3 years, and then annually for 5 years.

ELIGIBILITY:
1. Documentation of Disease

   A. Histologic Documentation:
   * Histologically documented mantle cell lymphoma with co-expression of CD20 (or CD19) and CD5 and lack of CD23 expression by immunophenotyping AND at least one of the following confirmatory tests:

     * positive immunostaining for cyclin D1; OR
     * the presence of t(11;14) on cytogenetic analysis; OR
     * molecular evidence of bcl-1/IgH rearrangement.
   * Cases that are CD5-negative and/or CD23-positive will be eligible provided that the histopathology is consistent with mantle cell lymphoma AND positive for cyclin D1, t(11;14), or bcl-1/IgH rearrangement.A tissue block should be submitted to the CALGB Pathology Coordinating Office for central pathology review.
   * A diagnosis based on peripheral blood or bone marrow is allowed. If the diagnosis is based only on blood, in addition to the immunophenotype and molecular confirmation above, a peripheral blood smear must be available for central pathology review. If the diagnosis is based on a bone marrow biopsy, the tissue block should be submitted.
   * Note: Failure to submit pathology materials within 60 days of patient registration will be considered a major protocol violation.

   B. Extent of Disease:
   * Stage I-IV. Patients with nodular histology mantle cell lymphoma must have Ann Arbor stage III or IV disease to be eligible. Patients with mantle zone histology will not be eligible because of their relatively favorable prognosis. Patients with other mantle cell histologies are eligible regardless of stage.
   * No active CNS disease defined as symptomatic meningeal lymphoma or known CNS parenchymal lymphoma. A lumbar puncture demonstrating mantle cell lymphoma at the time of registration to this study is not an exclusion for study enrollment.
2. Prior Treatment:

   A. Patients must be previously untreated or have received no more than one prior cycle of chemotherapy and/or rituximab treatment.

   B. No prior radiation therapy for mantle cell lymphoma.

   C. ≥ 2 weeks since major surgery.

   D. ≥ 3 weeks since prior chemotherapy.
3. Age Eligibility: Age ≥ 18 years and < 70 years
4. Murine Products Hypersensitivity Eligibility: No known hypersensitivity to murine products.
5. Use of Systemic Corticosteroids Eligibility: No medical condition requiring chronic use of systemic corticosteroids.
6. Eligibility Criteria on HIV Infection: No HIV infection. Patients with a history of intravenous drug abuse or any behavior associated with an increased risk of HIV infection should be tested for exposure to the HIV virus. Patients who test positive or who are known to be infected are not eligible due to an increased risk of infection with this regimen. An HIV test is not required for entry on this protocol, but is required if the patient is perceived to be at risk.
7. Non-pregnant and non-nursing: Non-pregnant and non-nursing. Treatment under this protocol would expose an unborn child to significant risks. Women and men of reproductive potential should agree to use an effective means of birth control.
8. HepBSAg or HepC Ab Eligibility: Patients who test positive for HepBSAg or HepC Ab are eligible provided all of the following criteria are met:

   A. bilirubin ≤ 2 x upper limit of normal; AND

   B. AST ≤ 3 x upper limit of normal; AND

   C. liver biopsy demonstrates ≤ grade 2 fibrosis and no cirrhosis.

   Hepatitis B surface Ag(+) patients will be treated with lamivudine (3TC) throughout protocol therapy and for 6-12 months thereafter.
9. Secondary Malignancy Eligibility: Patients with a "currently active" second malignancy, other than non-melanoma skin cancers are not eligible. This includes Waldenstrom's Macroglobulinemia, since such patents have experienced transient increases in IgM following initiation of rituximab, with the potential for hyperviscosity syndrome requiring plasmapheresis. Patients are not considered to have a "currently active" malignancy if they have completed anti-cancer therapy, and are considered by their physician to be at less than 30% risk of relapse.
10. Initial Required Laboratory Values:

    * LVEF by MUGA or ECHO ≥ 45%
    * Creatinine ≤ 2.0 mg/dL
    * Total Bilirubin ≤ 2.0 mg/dL (Unless attributable to Gilbert's Disease)
    * u-HCG or serum HCG Negative (If patient of childbearing potential).

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2006-06 (Actual); Primary Completion 2013-12 (Actual); Study Completion 2022-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence D. Kaplan, MD, Study Chair — University of California, San Francisco
Locations (48):
- United States (48):
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Illinois CancerCare - Bloomington, Bloomington, Illinois
  - St. Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital, Canton, Illinois
  - Illinois CancerCare - Canton, Canton, Illinois
  - Illinois CancerCare - Carthage, Carthage, Illinois
  - Memorial Hospital, Carthage, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Eureka Community Hospital, Eureka, Illinois
  - Illinois CancerCare - Eureka, Eureka, Illinois
  - Galesburg Clinic, PC, Galesburg, Illinois
  - Illinois CancerCare - Galesburg, Galesburg, Illinois
  - Illinois CancerCare - Havana, Havana, Illinois
  - Mason District Hospital, Havana, Illinois
  - Illinois CancerCare - Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare - Macomb, Macomb, Illinois
  - McDonough District Hospital, Macomb, Illinois
  - Illinois CancerCare - Monmouth, Monmouth, Illinois
  - OSF Holy Family Medical Center, Monmouth, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center, Normal, Illinois
  - Illinois CancerCare - Community Cancer Center, Normal, Illinois
  - Community Hospital of Ottawa, Ottawa, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Ottawa, Ottawa, Illinois
  - Illinois CancerCare - Pekin, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare - Peru, Peru, Illinois
  - Illinois Valley Community Hospital, Peru, Illinois
  - Illinois CancerCare - Princeton, Princeton, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - Illinois CancerCare - Spring Valley, Spring Valley, Illinois
  - Dana-Farber/Brigham and Women's Cancer Center, Boston, Massachusetts
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - Siteman Cancer Center at Barnes-Jewish Hospital - Saint Louis, St Louis, Missouri
  - Norris Cotton Cancer Center at Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Roswell Park Cancer Institute, Buffalo, New York
  - Monter Cancer Center of the North Shore-LIJ Health System, Lake Success, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - Don Monti Comprehensive Cancer Center at North Shore University Hospital, Manhasset, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Arthur G. James Cancer Hospital and Richard J. Solove Research Institute at Ohio State University Comprehensive Cancer Center, Columbus, Ohio

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From June 2006 to June 2010, 151 participants were enrolled at 14 sites and 147 participants received protocol treatment.
Pre-assignment Details: Of the 147 participants who began treatment, 102 participants were randomized. Participants who were not randomized are excluded from all analyses per study design.
Period: Overall Study
Arm/Group | Arm A Maintenance Therapy | Arm B Consolidation Therapy
Started | 52 | 50
Completed | 34 | 33
Not Completed | 18 | 17
Not completed — Adverse Event | 7 | 14
Not completed — Withdrawal by Subject | 4 | 3
Not completed — Progression | 6 | 0
Not completed — Non-protocol treatment | 1 | 0

BASELINE CHARACTERISTICS:
Population: 102 participants were randomized. Participants who were not randomized are excluded from all analyses per study design.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A Maintenance Therapy | Arm B Consolidation Therapy | Total
Number analyzed (Participants) | 52 | 50 | 102
Age, Continuous [Median (Full Range); unit: years] | 58 [29 to 69] | 59 [41 to 68] | 58.5 [29 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 12 | 22
  Male | 42 | 38 | 80
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 46 | 43 | 89
  Unknown or Not Reported | 6 | 6 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 0 | 3
  White | 46 | 48 | 94
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 2 | 5
Region of Enrollment [Number; unit: participants]
  United States | 52 | 50 | 102

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival Rate at 18 Months
Description: Progression free survival (PFS) rate at 18 months was defined as the proportion of patients that were alive and progression-free 18 months after registration into the study. The Kaplan-Meier method of 18 month progression-free survival was calculated..
Time Frame: At 18 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A Maintenance Therapy | Arm B Consolidation Therapy
Number analyzed (Participants) | 52 | 50
percentage of participants | 88.5 [80.2 to 97.6] | 96 [90.7 to 100]

2. Secondary Outcome: Overall Survival
Description: Overall Survival (OS) was measured from the date of study entry to date of death due to any cause. The median OS with 95% CI was estimated using the Kaplan-Meier method.
Time Frame: Up to 10 years
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | Arm A Maintenance Therapy | Arm B Consolidation Therapy
Number analyzed (Participants) | 52 | 50
years | NA [NA to NA] — The median, lower and upper limits for overall survival have not been reached. | 8.9 [7.2 to NA] — The upper limit was not calculable because an insufficient number of participants reached the event.

3. Secondary Outcome: Number of Participants With Complete Response Intensive Chemo-immunotherapy Plus Maintenance or Consolidation Bortezomib
Description: Complete response is:
  * Complete disappearance of all detectable clinical and radiographic evidence of target lesions and disappearance of all disease-related symptoms if present prior to therapy and normalization of biochemical abnormalities definitely assignable to NHL
  * All lymph nodes and nodal masses must have regressed to normal size (<= 1.5 cm in the greatest transverse diameter (GTD) for nodes > 1.5 cm prior to therapy) or <= 1 cm for nodes that were 1.1-1.5 cm in the GTD prior to therapy or by more than 75% in the sum of the products of the GTD
  * The spleen, if enlarged before therapy, must have regressed in size and must not be palpable on physical examination. Any macroscopic nodules in any organs detectable on imaging studies should no longer be present. Other organs enlarged prior to therapy due to involvement of lymphoma must have decreased in size
  * If bone marrow was involved by lymphoma prior to treatment, infiltrate must be cleared on repeat bone marrow aspirate
Time Frame: Up to 10 years
Measure: Number; unit: participants
Arm/Group | Arm A Maintenance Therapy | Arm B Consolidation Therapy
Number analyzed (Participants) | 52 | 80
participants | 31 | 35

4. Secondary Outcome: Number of Participants With Grade 3, 4 or 5 Adverse Event at Least Possibly Related to Treatment.
Description: The National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 3. Grade 1: Mild; Grade 2: Moderate; Grade 3: Severe; Grade 4: Life Threatening; Grade 5: Death.
Time Frame: Duration of treatment (up to approximately 2 years)
Measure: Number; unit: participants
Arm/Group | Arm A Maintenance Therapy | Arm B Consolidation Therapy
Number analyzed (Participants) | 52 | 50
participants | 52 | 50

ADVERSE EVENTS:
Arm/Group | Arm A Maintenance Therapy | Arm B Consolidation Therapy
Serious Adverse Events (participants affected / at risk) | 13/52 | 10/50
Other Adverse Events (participants affected / at risk) | 52/52 | 50/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A Maintenance Therapy (N=52) | Arm B Consolidation Therapy (N=50)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2) | 4 (4)
Hemoglobin decreased (Blood and lymphatic system disorders) | 10 (15) | 9 (10)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 2 (2)
Photophobia (Eye disorders) | 1 (1) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 1 (1)
Watering eyes (Eye disorders) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 5 (5) | 2 (2)
Colitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (3) | 1 (2)
Diarrhea (Gastrointestinal disorders) | 7 (8) | 4 (5)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 0 (0) | 2 (2)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gingival pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 3 (4) | 2 (2)
Nausea (Gastrointestinal disorders) | 7 (8) | 5 (7)
Oral pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 4 (5) | 3 (3)
Chest pain (General disorders) | 0 (0) | 1 (1)
Chills (General disorders) | 3 (3) | 3 (3)
Edema limbs (General disorders) | 3 (3) | 2 (2)
Fatigue (General disorders) | 8 (8) | 5 (5)
Fever (General disorders) | 3 (3) | 4 (4)
Pain (General disorders) | 2 (2) | 1 (1)
Cytokine release syndrome (Immune system disorders) | 2 (2) | 2 (2)
Hypersensitivity (Immune system disorders) | 1 (1) | 3 (3)
Catheter related infection (Infections and infestations) | 1 (1) | 1 (1)
Colitis, infectious (e.g., Clostridium difficile) (Infections and infestations) | 1 (2) | 0 (0)
Infectious colitis (Infections and infestations) | 0 (0) | 1 (1)
Infectious meningitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 3 (3) | 2 (2)
Skin infection (Infections and infestations) | 1 (1) | 0 (0)
Ureteritis (Infections and infestations) | 0 (0) | 1 (1)
Vascular access complication (Injury, poisoning and procedural complications) | 1 (1) | 1 (2)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1) | 3 (4)
Alanine aminotransferase increased (Investigations) | 5 (7) | 3 (3)
Alkaline phosphatase increased (Investigations) | 3 (3) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 7 (7) | 3 (3)
Blood bilirubin increased (Investigations) | 4 (4) | 4 (4)
Creatinine increased (Investigations) | 4 (4) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 0 (0)
INR increased (Investigations) | 0 (0) | 3 (4)
Leukocyte count decreased (Investigations) | 8 (11) | 6 (7)
Lymphocyte count decreased (Investigations) | 8 (10) | 9 (9)
Neutrophil count decreased (Investigations) | 10 (12) | 7 (9)
Platelet count decreased (Investigations) | 11 (15) | 9 (11)
Weight loss (Investigations) | 2 (2) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 4 (5) | 5 (5)
Blood glucose increased (Metabolism and nutrition disorders) | 6 (7) | 5 (6)
Blood uric acid increased (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Serum albumin decreased (Metabolism and nutrition disorders) | 5 (5) | 4 (5)
Serum calcium decreased (Metabolism and nutrition disorders) | 7 (8) | 5 (6)
Serum calcium increased (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Serum glucose decreased (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Serum magnesium decreased (Metabolism and nutrition disorders) | 1 (2) | 2 (2)
Serum phosphate decreased (Metabolism and nutrition disorders) | 0 (0) | 4 (4)
Serum potassium decreased (Metabolism and nutrition disorders) | 4 (5) | 5 (6)
Serum sodium decreased (Metabolism and nutrition disorders) | 6 (6) | 3 (3)
Serum sodium increased (Metabolism and nutrition disorders) | 0 (0) | 2 (3)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ataxia (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 3 (3)
Headache (Nervous system disorders) | 5 (5) | 3 (5)
Hydrocephalus (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 4 (5) | 2 (2)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 3 (4) | 0 (0)
Confusion (Psychiatric disorders) | 0 (0) | 3 (3)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (2) | 2 (2)
Urogenital disorder (Renal and urinary disorders) | 0 (0) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Hand-and-foot syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash desquamating (Skin and subcutaneous tissue disorders) | 4 (4) | 2 (2)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Sweating (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 3 (3) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A Maintenance Therapy (N=52) | Arm B Consolidation Therapy (N=50)
Febrile neutropenia (Blood and lymphatic system disorders) | 32 (46) | 27 (43)
Hemoglobin decreased (Blood and lymphatic system disorders) | 38 (357) | 44 (307)
Hemolysis (Blood and lymphatic system disorders) | 3 (3) | 3 (7)
Lymph node pain (Blood and lymphatic system disorders) | 0 (0) | 3 (3)
Lymphatic disorder (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Transfusion: Platelets (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
Transfusion: pRBCs (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
Arrhythmia supraventricular (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 4 (4) | 3 (5)
Atrial flutter (Cardiac disorders) | 1 (1) | 1 (1)
Atrial tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Atrioventricular block first degree (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac disorder (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac pain (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac valve disease (Cardiac disorders) | 1 (1) | 2 (2)
Conduction disorder (Cardiac disorders) | 0 (0) | 1 (1)
Edema (Cardiac disorders) | 3 (5) | 1 (2)
Left ventricular failure (Cardiac disorders) | 3 (3) | 1 (1)
Palpitations (Cardiac disorders) | 3 (4) | 3 (12)
Pericardial effusion (Cardiac disorders) | 0 (0) | 2 (2)
Pericarditis (Cardiac disorders) | 1 (1) | 0 (0)
Sinus arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 3 (5) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 8 (9) | 6 (7)
Supraventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (2)
Supraventricular tachycardia (Cardiac disorders) | 2 (3) | 2 (2)
Ventricular arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Ear disorder (Ear and labyrinth disorders) | 0 (0) | 2 (2)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 1 (2)
External ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Hearing impaired (Ear and labyrinth disorders) | 3 (4) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Conjunctivitis (Eye disorders) | 1 (1) | 0 (0)
Diplopia (Eye disorders) | 0 (0) | 1 (1)
Dry eye syndrome (Eye disorders) | 4 (8) | 4 (6)
Extraocular muscle paresis (Eye disorders) | 0 (0) | 2 (5)
Eye disorder (Eye disorders) | 4 (6) | 2 (2)
Eye pain (Eye disorders) | 1 (1) | 2 (2)
Photophobia (Eye disorders) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 7 (11) | 3 (4)
Watering eyes (Eye disorders) | 3 (3) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 6 (10) | 2 (3)
Abdominal pain (Gastrointestinal disorders) | 16 (32) | 18 (29)
Anal pain (Gastrointestinal disorders) | 0 (0) | 2 (2)
Colitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Colonic hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 28 (59) | 28 (70)
Diarrhea (Gastrointestinal disorders) | 45 (144) | 45 (124)
Dry mouth (Gastrointestinal disorders) | 2 (2) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 12 (14) | 9 (17)
Dysphagia (Gastrointestinal disorders) | 5 (7) | 8 (9)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 5 (5) | 7 (13)
Enteritis (Gastrointestinal disorders) | 3 (3) | 0 (0)
Esophageal pain (Gastrointestinal disorders) | 3 (4) | 5 (5)
Esophagitis (Gastrointestinal disorders) | 1 (1) | 2 (3)
Flatulence (Gastrointestinal disorders) | 5 (8) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastrointestinal disorder (Gastrointestinal disorders) | 4 (6) | 1 (1)
Gingival pain (Gastrointestinal disorders) | 1 (2) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 7 (8) | 6 (7)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 35 (52) | 35 (58)
Nausea (Gastrointestinal disorders) | 47 (170) | 48 (170)
Oesophagoscopy abnormal (Gastrointestinal disorders) | 0 (0) | 1 (2)
Oral hemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0)
Oral pain (Gastrointestinal disorders) | 1 (3) | 3 (4)
Peritoneal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Proctitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2)
Rectal pain (Gastrointestinal disorders) | 2 (2) | 5 (6)
Salivary gland disorder (Gastrointestinal disorders) | 1 (1) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 2 (2) | 2 (2)
Toothache (Gastrointestinal disorders) | 1 (1) | 2 (2)
Typhlitis (Gastrointestinal disorders) | 2 (2) | 1 (1)
Vomiting (Gastrointestinal disorders) | 45 (103) | 44 (95)
Chest pain (General disorders) | 4 (4) | 6 (7)
Chills (General disorders) | 24 (36) | 25 (48)
Death NOS (General disorders) | 0 (0) | 1 (1)
Edema limbs (General disorders) | 16 (42) | 18 (36)
Facial pain (General disorders) | 0 (0) | 1 (4)
Fatigue (General disorders) | 44 (284) | 45 (257)
Fever (General disorders) | 28 (47) | 26 (37)
Flu-like symptoms (General disorders) | 2 (4) | 0 (0)
Gait abnormal (General disorders) | 1 (1) | 0 (0)
General symptom (General disorders) | 1 (1) | 1 (2)
Hypothermia (General disorders) | 1 (1) | 0 (0)
Ill-defined disorder (General disorders) | 1 (1) | 1 (1)
Localized edema (General disorders) | 5 (5) | 5 (6)
Pain (General disorders) | 14 (24) | 10 (15)
Radiation-Other(Specify,_____) (General disorders) | 0 (0) | 1 (1)
Hepatobiliary disease (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cytokine release syndrome (Immune system disorders) | 6 (7) | 10 (13)
Hypersensitivity (Immune system disorders) | 7 (11) | 11 (15)
Serum sickness (Immune system disorders) | 1 (1) | 0 (0)
Abdominal infection (Infections and infestations) | 2 (2) | 1 (1)
Anal infection (Infections and infestations) | 0 (0) | 1 (1)
Anorectal infection (Infections and infestations) | 0 (0) | 1 (1)
Arteritis infective (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 4 (5) | 0 (0)
Catheter related infection (Infections and infestations) | 9 (12) | 12 (15)
Colitis, infectious (e.g., Clostridium difficile) (Infections and infestations) | 2 (3) | 1 (2)
Conjunctivitis infective (Infections and infestations) | 0 (0) | 2 (3)
Gingival infection (Infections and infestations) | 3 (5) | 2 (2)
Infection (Infections and infestations) | 4 (4) | 6 (9)
Infection with grade 3 or 4 neutropenia (Infections and infestations) | 0 (0) | 2 (3)
Infection without neutropenia (Infections and infestations) | 0 (0) | 2 (2)
Infectious colitis (Infections and infestations) | 4 (4) | 2 (2)
Lip infection (Infections and infestations) | 2 (2) | 1 (1)
Mucosal infection (Infections and infestations) | 1 (1) | 0 (0)
Nail infection (Infections and infestations) | 1 (1) | 0 (0)
Opportunistic infection (Infections and infestations) | 0 (0) | 2 (2)
Otitis externa (Infections and infestations) | 1 (2) | 0 (0)
Otitis media (Infections and infestations) | 2 (2) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 8 (12) | 5 (8)
Rhinitis infective (Infections and infestations) | 3 (3) | 1 (1)
Sepsis (Infections and infestations) | 7 (7) | 5 (6)
Sinusitis (Infections and infestations) | 11 (11) | 6 (8)
Skin infection (Infections and infestations) | 4 (4) | 7 (12)
Tooth infection (Infections and infestations) | 1 (2) | 1 (1)
Tracheitis (Infections and infestations) | 1 (1) | 0 (0)
Upper aerodigestive tract infection (Infections and infestations) | 1 (1) | 1 (1)
Upper respiratory infection (Infections and infestations) | 14 (19) | 6 (6)
Ureteritis (Infections and infestations) | 2 (3) | 2 (2)
Urinary tract infection (Infections and infestations) | 5 (5) | 3 (6)
Vaginal infection (Infections and infestations) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 3 (3) | 3 (3)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Gastrointestinal anastomotic leak (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Intraoperative neurological injury - Spinal cord (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular access complication (Injury, poisoning and procedural complications) | 3 (4) | 4 (4)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 6 (12) | 7 (9)
Alanine aminotransferase increased (Investigations) | 26 (99) | 27 (86)
Alkaline phosphatase (Investigations) | 1 (1) | 1 (1)
Alkaline phosphatase increased (Investigations) | 17 (32) | 19 (56)
Aspartate aminotransferase increased (Investigations) | 29 (92) | 31 (95)
Blood bilirubin increased (Investigations) | 15 (33) | 16 (54)
CD4 lymphocytes decreased (Investigations) | 1 (1) | 3 (3)
Cardiac troponin T increased (Investigations) | 1 (1) | 1 (1)
Creatinine increased (Investigations) | 11 (25) | 11 (27)
Fibrinogen decreased (Investigations) | 0 (0) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 4 (11) | 1 (3)
INR increased (Investigations) | 7 (13) | 5 (7)
Laboratory test abnormal (Investigations) | 1 (2) | 2 (2)
Leukocyte count decreased (Investigations) | 37 (261) | 38 (229)
Leukocytes (total WBC) for BMT studies, if specified in the protocol. (Investigations) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 35 (285) | 38 (264)
Neutrophil count decreased (Investigations) | 52 (283) | 50 (300)
Platelet count decreased (Investigations) | 52 (472) | 50 (399)
Serum cholesterol increased (Investigations) | 0 (0) | 1 (1)
Weight gain (Investigations) | 10 (15) | 9 (10)
Weight loss (Investigations) | 10 (18) | 12 (15)
Acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 32 (55) | 35 (83)
Blood glucose increased (Metabolism and nutrition disorders) | 27 (217) | 23 (135)
Blood uric acid increased (Metabolism and nutrition disorders) | 4 (4) | 3 (4)
Dehydration (Metabolism and nutrition disorders) | 7 (8) | 8 (13)
Glucose intolerance (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Serum albumin decreased (Metabolism and nutrition disorders) | 22 (57) | 23 (60)
Serum calcium decreased (Metabolism and nutrition disorders) | 29 (126) | 25 (85)
Serum calcium increased (Metabolism and nutrition disorders) | 3 (3) | 4 (8)
Serum glucose decreased (Metabolism and nutrition disorders) | 9 (14) | 9 (17)
Serum magnesium decreased (Metabolism and nutrition disorders) | 15 (29) | 13 (28)
Serum magnesium increased (Metabolism and nutrition disorders) | 6 (7) | 8 (12)
Serum phosphate decreased (Metabolism and nutrition disorders) | 15 (25) | 11 (20)
Serum potassium decreased (Metabolism and nutrition disorders) | 28 (80) | 22 (67)
Serum potassium increased (Metabolism and nutrition disorders) | 4 (7) | 7 (10)
Serum sodium decreased (Metabolism and nutrition disorders) | 24 (73) | 21 (71)
Serum sodium increased (Metabolism and nutrition disorders) | 10 (17) | 8 (10)
Serum triglycerides increased (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 16 (48) | 15 (33)
Arthritis (Musculoskeletal and connective tissue disorders) | 3 (13) | 2 (8)
Back pain (Musculoskeletal and connective tissue disorders) | 15 (36) | 13 (20)
Bone pain (Musculoskeletal and connective tissue disorders) | 14 (25) | 8 (12)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 5 (6) | 4 (4)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 5 (15) | 12 (22)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (5)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 7 (11) | 3 (8)
Myalgia (Musculoskeletal and connective tissue disorders) | 11 (29) | 12 (28)
Neck pain (Musculoskeletal and connective tissue disorders) | 7 (16) | 6 (6)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (5)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 16 (29) | 12 (19)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Acoustic nerve disorder NOS (Nervous system disorders) | 1 (1) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 1 (1)
Cognitive disturbance (Nervous system disorders) | 2 (2) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 16 (24) | 14 (17)
Dysgeusia (Nervous system disorders) | 8 (12) | 9 (12)
Extrapyramidal disorder (Nervous system disorders) | 3 (7) | 1 (1)
Facial muscle weakness (Nervous system disorders) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 32 (85) | 33 (56)
Hydrocephalus (Nervous system disorders) | 0 (0) | 1 (1)
Ischemia cerebrovascular (Nervous system disorders) | 2 (2) | 1 (1)
Memory impairment (Nervous system disorders) | 7 (11) | 2 (4)
Neuralgia (Nervous system disorders) | 6 (27) | 10 (26)
Neurological disorder NOS (Nervous system disorders) | 4 (5) | 1 (3)
Nystagmus (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 11 (37) | 4 (11)
Peripheral sensory neuropathy (Nervous system disorders) | 38 (243) | 42 (216)
Phrenic nerve paralysis (Nervous system disorders) | 0 (0) | 2 (4)
Radiculitis brachial (Nervous system disorders) | 0 (0) | 2 (4)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Sinus pain (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 6 (7) | 2 (4)
Syncope vasovagal (Nervous system disorders) | 0 (0) | 2 (2)
Tremor (Nervous system disorders) | 2 (2) | 4 (5)
Agitation (Psychiatric disorders) | 0 (0) | 1 (3)
Anxiety (Psychiatric disorders) | 13 (38) | 14 (24)
Confusion (Psychiatric disorders) | 1 (1) | 4 (7)
Depression (Psychiatric disorders) | 3 (4) | 10 (17)
Insomnia (Psychiatric disorders) | 19 (50) | 29 (74)
Libido decreased (Psychiatric disorders) | 1 (1) | 1 (1)
Psychosis (Psychiatric disorders) | 0 (0) | 1 (1)
Bladder hemorrhage (Renal and urinary disorders) | 1 (1) | 2 (2)
Bladder pain (Renal and urinary disorders) | 1 (1) | 1 (1)
Glomerular filtration rate decreased (Renal and urinary disorders) | 2 (2) | 0 (0)
Hemoglobin urine positive (Renal and urinary disorders) | 1 (2) | 0 (0)
Proteinuria (Renal and urinary disorders) | 2 (3) | 1 (1)
Urethral pain (Renal and urinary disorders) | 1 (2) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 1 (1) | 8 (10)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 2 (3)
Urinary retention (Renal and urinary disorders) | 0 (0) | 4 (5)
Urine discoloration (Renal and urinary disorders) | 1 (1) | 0 (0)
Urogenital disorder (Renal and urinary disorders) | 3 (7) | 1 (3)
Breast pain (Reproductive system and breast disorders) | 2 (2) | 1 (2)
Erectile dysfunction (Reproductive system and breast disorders) | 2 (2) | 1 (1)
Gynecomastia (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Pelvic floor muscle weakness (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Scrotal pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Testicular pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vaginal hemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 17 (30) | 10 (15)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 30 (64) | 18 (33)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 22 (53) | 19 (55)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 11 (14)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 3 (5)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (3)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 10 (10)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (6) | 1 (3)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 12 (22)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 1 (1)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 2 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 19 (30) | 5 (10)
Dry skin (Skin and subcutaneous tissue disorders) | 5 (5) | 4 (5)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)
Hand-and-foot syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Nail disorder (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (2)
Pain of skin (Skin and subcutaneous tissue disorders) | 4 (8) | 2 (2)
Petechiae (Skin and subcutaneous tissue disorders) | 3 (3) | 5 (5)
Photosensitivity (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 9 (14) | 9 (12)
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0)
Rash desquamating (Skin and subcutaneous tissue disorders) | 34 (62) | 31 (73)
Skin disorder (Skin and subcutaneous tissue disorders) | 7 (10) | 7 (11)
Skin induration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Sweating (Skin and subcutaneous tissue disorders) | 11 (23) | 12 (17)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (3) | 2 (3)
Flushing (Vascular disorders) | 7 (8) | 7 (8)
Hemorrhage (Vascular disorders) | 2 (2) | 1 (1)
Hot flashes (Vascular disorders) | 0 (0) | 2 (2)
Hypertension (Vascular disorders) | 5 (12) | 12 (15)
Hypotension (Vascular disorders) | 13 (18) | 15 (19)
Phlebitis (Vascular disorders) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 5 (6) | 1 (1)
Vasculitis (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less